CLINICAL TRIAL: NCT05312827
Title: Training Intervention and Program of Support (TIPS) for Fostering the Adoption of Family-centred Telehealth Interventions in Pediatric Rehabilitation: A Pan-Canadian Implementation-effectiveness Study
Brief Title: Training Intervention and Program of Support (TIPS): Fostering Family-centred Telehealth in Pediatric Rehabilitation
Acronym: TIPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Chantal Camden, Dr. Chantal Camden, Université de Sherbrooke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022-4546
Record Dates: First submitted 2022-02-15; First posted 2022-04-06 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Telerehabilitation
Keywords: telehealth; family-centred; pediatric rehabilitation
MeSH Terms: interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Intervention Model Description: A 4-year pan-Canadian stakeholder-oriented, mixed-method implementation-effectiveness design will be used. TIPS will be implemented in all sites in a same region during the same month, and sequentially introduced across all regions, 2 months apart. An interrupted time series (ITS) was selected to assess primary implementation outcomes (obj. 1), as recommended for research in real-world settings. An ITS consists of observing the same dependent variables over time, with a break in the series of observations corresponding to the introduction of an intervention. If the intervention is effective, a change in the series' pre- and post-intervention averages will be observed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telehealth (Experimental): The proposed pre-post study will evaluate the implementation and effectiveness of a Training Intervention and Program of Support (TIPS) to enhance the adoption of family-centred telehealth in pediatric rehabilitation centres across Canada. TIPS is a multifaceted intervention, comprised of the following: 1) a 10-hour intensive training program offered to participating therapists at each site over a one-month period, including 4 hours of self-paced learning modules and a 6-hour mandatory interactive webinar; and 2) an 11-month program of support which is composed of monthly mentoring meetings at each site led by the local therapist champion, and a national virtual community of practice facilitated by 3 national knowledge brokers - an occupational therapist, a physiotherapist and a speech-language pathologist - experienced in family-centred telehealth in pediatric rehabilitation, offered simultaneously to all participating therapists across Canada.
  Interventions: Behavioral: Training Intervention and Program of Support (TIPS) for fostering the adoption of family-centred telehealth interventions in pediatric rehabilitation

INTERVENTIONS:
Behavioral: Training Intervention and Program of Support (TIPS) for fostering the adoption of family-centred telehealth interventions in pediatric rehabilitation — The proposed pre-post study will evaluate the implementation and effectiveness of a Training Intervention and Program of Support (TIPS) to enhance the adoption of family-centred telehealth in pediatric rehabilitation centres across Canada. TIPS is a multifaceted intervention, comprised of the following: 1) a 10-hour intensive training program offered to participating therapists at each site over a one-month period, including 4 hours of self-paced learning modules and a 6-hour mandatory interactive webinar; and 2) an 11-month program of support which is composed of monthly mentoring meetings at each site led by the local therapist champion, and a national virtual community of practice facilitated by 3 national knowledge brokers - an occupational therapist, a physiotherapist and a speech-language pathologist - experienced in family-centred telehealth in pediatric rehabilitation, offered simultaneously to all participating therapists across Canada.
  Other Names: TIPS

SUMMARY:
Timely access to family-centred services for children with disability and their families is important to support their development and well-being. Currently, many children face long wait times and barriers to services. Lack of access can lead to negative impacts for children and stress for their families. With the COVID-19 pandemic, these issues have been made more challenging with the loss of rehabilitation support for children, increasing stress on families. During this time, therapists moved to telehealth service delivery to support children and families.

We know that telehealth can improve access to services, children's outcomes, and family satisfaction, and that telehealth a key element of Family Centred Services (FCS) in pediatric rehabilitation. FCC include practices that promote flexibility, respect and dignity for families' views, knowledge and strengths, effective information sharing, partnership and collaboration in decision making, and coordinated and comprehensive care. FCC focuses on developing collaborative family-provider relationships, where parents are active participants in collaborative goal-setting, therapy planning, implementation, and evaluation, and where activities are integrated within daily routines and contexts (e.g., home and community). Compared to traditional service delivery methods, telehealth offers opportunities to enhance FCC practices. FCC provides alternate, convenient, and flexible ways to partner with families, respecting their characteristics and barriers, allows knowledge and information sharing about the child within their contexts, supports family decision making and parents' well-being, and has been recognized as an important addition to comprehensive care coordination and service delivery.

Telehealth is an important and effective alternative for families living in both urban and remote or underserved areas and can be more convenient than in-person visits (e.g., less travel time, schedule flexibility). However, the use of telehealth prior to the pandemic was low in pediatric rehabilitation. In addition, many therapists report delivering telehealth without prior experience, and lack confidence, knowledge, and training in effective intervention strategies. Although therapists' knowledge, skills and attitudes toward telehealth can improve with time and experience, training and support are required for behavioural changes to occur.

Following the pandemic, there has been continued support for the use of FCT and for its ongoing use to support families of children with disability. Pediatric rehabilitation therapists, service managers, professional associations, policy makers, and families are all making the case for not "returning to normal", and are asking for help to keep telehealth as part of FCS care.

The goal of the current study is to evaluate the use and effectiveness of a Training Intervention and Program of Support (TIPS) to increase the uptake of FCT in pediatric rehabilitation centres across Canada.

The main research question is: Can TIPS be adapted to increase the use of FCT interventions by therapists working in different contexts?

The primary objectives are to:

1. Evaluate the use of FCT regarding:

   1. Therapists' desire to use vs actual use of FCT practices
   2. Use of FCT practices as they were intended to be used

   Secondary objectives are to:
2. Describe the variations required to adapt the TIPS to meet each site's needs
3. Identify factors that influence FCT use and adherence
4. Evaluate the effectiveness with regards to:

   1. Service wait-times
   2. Family-centredness of services
   3. Changes in service delivery
5. Evaluate the costs (and possible cost savings) related to increased use of FCT

The primary hypotheses are that therapists' desire to adopt FCT and deliver FCT practices as intended will (i) improve slightly in the short term (i.e., one-month post-TIPS), yet (ii) will improve significantly post-TIPS, (iii) while actual use will vary over time, across sites and therapists, and will depend on therapist-, client-, organizational- and system-factors. For the secondary hypotheses, the investigators expect that, for sites with the largest changes in desire to use and use of FCT practices as intended, (iv) wait times will significantly decrease and (v) families' perceptions of service quality will significantly improve post-TIPS.

DETAILED DESCRIPTION:
INTRODUCTION Timely access to family-centred services for children with disability and their families is crucial to support their development and well-being. Currently, many children face long wait times (i.e., up to 2 years) and organizational, geographic and/or cultural barriers to services. Lack of access can lead to negative developmental, health and social consequences for children (e.g., suboptimal development, academic difficulties) and their families (e.g., stress). The COVID-19 pandemic further exacerbated these issues, as rehabilitation support for children was lost, increasing parental mental health burden (e.g., increased stress, depression). To minimize the negative impacts of these service disruptions, therapists were required to shift to telehealth service delivery.

Evidence exists of the efficacy of telehealth to improve service access, children's outcomes, and family satisfaction and acceptability, supporting the integration of telehealth as a key element of Family Centred Services (FCS) in pediatric rehabilitation. Telehealth can be defined as 'any asynchronous or real time clinical intervention provided remotely by therapists to patients and/or caregivers. It has been recognized as an important alternative for families living in underserved or remote areas. However, some families in well-served urban locations also prefer the convenience of telehealth over in-person visits (e.g., less travel time, schedule flexibility). Prior to the pandemic, a systematic review of pediatric rehabilitation telehealth randomized controlled trials supported the efficacy of such interventions for a wide range of outcomes and diverse populations. Further publications demonstrated the efficacy and acceptability of telehealth, further supporting its integration into comprehensive FCS models.

The established efficacy of telehealth highlights a critical knowledge-to-practice gap. Before the pandemic, the adoption of telehealth was low in pediatric rehabilitation. In an international survey conducted in August 2019 (1,133 pediatric therapists from 76 countries), 3.9% were using telehealth; a follow-up survey with a subsample in May 2020 highlighted that 70.1% had adopted telehealth. Many reported doing so without prior experience, and lacked confidence, knowledge, and training in effective intervention strategies. When asked what support was required to implement telehealth, training was by far the most frequently cited - and included communication skills with families over the phone and internet, safe and effective use of platforms, reliable assessment, and intervention strategies with children of various ages and health conditions. Although therapists' knowledge, skills and attitudes toward telehealth can improve with time and experience, training and support are required for behavioural changes to occur. Unfortunately, there is a paucity of evidence related to how personal and contextual factors may influence telehealth training and support. Targeting therapists' knowledge, skills, and attitudes, associated with their intention to adopt telehealth, and their professional role within FCS, appear vital to the implementation of telehealth.

For the purposes of this study, family-centred telehealth (FCT) is defined as pediatric rehabilitation which uses family-centred care (FCC) practices while working with families remotely. FCC is recognized as a best practice approach in pediatric rehabilitation. Described as a partnership approach, FCC is based on the belief that the child's well-being and care needs are best supported within the family context through effective family-provider collaborations. Moreover, FCC's central tenet is the assumption that the processes of care delivery are as important to the child and family outcomes as the specific characteristic of the clinical intervention delivered. It is characterized by practices that promote clinical flexibility, respect and dignity for families' perspectives, knowledge, strengths and characteristics, effective information sharing (general and specific), partnership and collaboration between parties to support decision making, and coordinated and comprehensive care delivery. Furthermore, FCC occurs in the therapeutic environment that optimizes the development of a collaborative family-provider relationship, where parents are active participants in collaborative goal-setting, therapy planning, implementation, and evaluation, and where activities are integrated within daily routines and contexts (e.g., home and community). Compared to more traditional service delivery methods, telehealth offers opportunities to enhance FCC practices. It provides alternate, convenient, and flexible ways to partner with families, respecting their characteristics (e.g., single parenting) and constraints (e.g., geographical, temporal, financial), allows real-time knowledge acquisition and information sharing about the child within their contexts, supports family decision making and parents' psychosocial well-being (i.e., decreasing anxiety, stress, and depression), and has been recognized as an important addition to comprehensive care coordination and service delivery.

Considerable momentum exists supporting the uptake of FCT and fostering its ongoing sustainable use within accessible and supportive services for the families of children with disability following the pandemic. Pediatric rehabilitation therapists, service managers, professional associations, policy makers, and patients alike are calling for resistance to "returning to normal", and instead are requesting help to sustain telehealth as part of the FCS continuum of care. The proposed study aims to evaluate the implementation and effectiveness of a Training Intervention and Program of Support (TIPS) to enhance the adoption of FCT in pediatric rehabilitation centres across Canada.

RESEARCH QUESTIONS AND OBJECTIVES The main research question is: Can TIPS be co-adapted to enhance the adoption of FCT interventions by therapists working in different contexts?

Primary objectives are to:

1. Evaluate the implementation with regard to:

   1. Therapists' intention to adopt vs actual adoption of FCT practices
   2. Fidelity of FCT practices

   Secondary objectives are to:
2. Document the contextual variations required to co-adapt the TIPS to meet each site's needs
3. Identify factors influencing FCT adoption and fidelity
4. Evaluate the effectiveness with regards to:

   1. Service wait-times
   2. Families' perception of service quality (i.e., family-centredness)
   3. Changes in service delivery
5. Evaluate the costs (and possible cost savings) related to increased use of FCT

The primary hypotheses are that therapists' intention to adopt FCT and fidelity of FCT practices will (i) improve minimally in the short term (i.e., one-month post-TIPS), yet (ii) will improve significantly post-implementation of TIPS, (iii) while actual adoption and engagement will fluctuate over time, across sites and therapists, and will depend on therapist-, client-, organizational- and system-factors. For the secondary hypotheses, the investigators expect that, for sites with the largest effect change in intention to adopt and fidelity of FCT practices, (iv) wait times will significantly decrease and (v) families' perceptions of service quality will significantly improve post-implementation of TIPS.

METHODS Implementation science conceptual framework The study framework builds on implementation science frameworks that aim to accelerate the translational research pipeline, bridging the current knowledge-to-practice gap. Specifically, the Consolidated Framework for Implementation Research (CFIR) will guide the identification of factors influencing adoption of FCT and will help engage leaders in participating sites in adapting the TIPS to their own contextual drivers, while maintaining the FCT key ingredients. A hybrid design will be used, as recommended when the traditional research pipeline efficacy-effectiveness-implementation is too time consuming, and considered unethical, failing to adequately respond to the urgency of the expressed need. A Type 3 hybrid design was chosen, primarily focusing on implementation indicators, while also collecting some effectiveness outcomes, with comparative assessments occurring at the therapist, service and/or family level. This design is recommended when there is: 1) momentum for implementation within the health care system; 2) strong face validity and indirect evidence for the clinical intervention and implementation strategy to support generalizability; 3) minimal risk associated with the clinical intervention and the implementation strategy; and 4) evidence of feasibility for the implementation strategy and support in the clinical and organization context under study. The present study meets all these criteria, as there is: 1) momentum for the sustainability of telehealth implemented during and following the COVID-19 pandemic; 2) strong and growing evidence of effectiveness for telehealth, as well as for training and support knowledge translation strategies; 3) promising results from our studies supporting the safe use of TIPS to implement FCT; and 4) well-established evidence of implementation feasibility of telehealth.

Design A 4-year pan-Canadian stakeholder-oriented, mixed-method implementation-effectiveness design will be used. TIPS will be implemented in all sites in a same region during the same month, and sequentially introduced across all regions, 2 months apart. An interrupted time series (ITS) was selected to assess primary implementation outcomes (obj. 1), as recommended for research in real-world settings. An ITS consists of observing the same dependent variables over time, with a break in the series of observations corresponding to the introduction of an intervention. If the intervention is effective, a change in the series' pre- and post-intervention averages will be observed.

Intervention Informed by implementation strategies recognized as effective in pediatric rehabilitation, TIPS is a multifaceted intervention, comprised of the following components: 1) a 10-hour intensive training program offered to participating therapists at each site over a one-month period, which includes 4 hours of self-paced learning modules and a 6-hour mandatory interactive webinar; and 2) an 11-month program of support which is composed of monthly mentoring meetings at each site led by the local therapist champion, and a national virtual community of practice (vCoP) facilitated by 3 national knowledge brokers (KBs) - an occupational therapist (OT), a physiotherapist (PT) and a speech-language pathologist (SLP) - experienced in FCT in pediatric rehabilitation, offered simultaneously to all participating therapists across Canada.

The TIPS self-paced learning modules are informed by contemporary frameworks of FCC, and relevant family-oriented services. More specifically, they will address the key ingredients associated with the FCT processes and provide practice examples. These key ingredients include: 1) service operations (e.g., service coordination, organization and structures, care planning and goal setting), 2) participatory (e.g., parent engagement, focus on individual family's needs) and 3) relational (e.g., active listening, respect, empathy, reciprocity) caregiving, 4) communicating general (e.g., access to current and future services, parent groups) and specific (e.g., co-morbidities associated with child's condition) information, as well as 6) coaching (e.g., parent task analysis, caregiver implemented strategies with natural contexts, solution-focused coaching)., and 7) engagement strategies. Multimedia (e.g., videos, presentations) content for the asynchronous training modules will be developed by several members of the study team, through ongoing consultation with experts in the field, using education course creation software. The curriculum will then be uploaded to a password protected online platform, for which a unique username and password will be required. Knowledge acquisition, based on the specified learning objectives and the key messages targeted in each training module, will be assessed through short pedagogical quizzes. Completion of the asynchronous modular training and knowledge assessment will be recommended prior to undertaking the synchronous webinar(s).

A 6-hour synchronous webinar component will also be delivered by members of the research team and the 3 national KBs. These webinars will engage therapists in discussion (e.g., case studies), interactive activities (e.g., role play, simulations) to build their critical thinking on how to implement these practices in their context. The webinar content will be adapted for each site in consultation with the Local Leadership Team, (i.e., the site manager, a therapist champion, and a parent/patient partner). This co-adaptation phase will ensure content is tailored to individual site contexts (e.g., engagement practices, site clinical goal-setting processes, service coordination as per team procedures), learner-centred and clinically relevant. The FCT interventions can be implemented using a variety of technologies, including various videoconferencing options, online platforms, websites, email systems, and even telephone. Therapists will be encouraged to consider various asynchronous and real-time technologies, which best respond to families' needs and preferences, and those approved by their organizations. The research team will refrain from recommending specific technologies. There is no prescribed frequency or duration for the FCT interventions; therapist participants will work with families according to their goals and preferences, and organizational policies.

Finally, a program of support will be offered for the remaining year via monthly videoconference mentoring meetings, and access to the vCoP also housed on the password-protected platform. Monthly meetings will focus on sharing site-specific successes, challenges, proposing solutions and reporting results, as well as sharing useful and practical resources. The vCoP will be used to canvas for solutions to address challenges at a national level, share successes, discuss specific cases for guidance, feedback and input, and to share useful tips and tricks, and resources. The structure of our vCoP was informed by previous work related to vCoP and KBs (i.e., individuals with content and leadership expertise, who foster information sharing and research evidence use).

Study Settings Participating sites are publicly funded organizations providing outpatient pediatric rehabilitation services to children aged 0-12 years with or at risk of disability. 'Disability' is used inclusively to recognize all medical diagnoses resulting in limitations in function, such as cerebral palsy and autism spectrum disorder. The term "at risk" includes children presenting with delayed development who may not yet have a diagnosis but have clear functional limitations and qualify for rehabilitation services. The upper age limit of 12 years was chosen, as best practices regarding transition of care suggest that different relationships should be fostered with adolescents over 12 years. The 20 participating sites selected based on various characteristics (e.g., populations, size, services provided, catchment area) thought to influence outcomes, the effect of which will be explored, are clustered into 6 provincial regions. TIPS will be sequentially introduced (i.e., 2 months apart) to each of the regions. To limit the risk of contamination, TIPS will be introduced to all sites in the same region in the same month. However, training will be conducted on a site-by-site basis to create team cohesion. The 2-month interval for implementation between regions gives flexibility for organizing implementation and data collection activities based on site availability and vacation schedules.

Study participants

Participants will belong to at least one of the following categories:

1. Managers (n=20, one per site): Person responsible for rehabilitation services at the site, or their delegate. The managers were identified during the selection of study sites. As members of the Local Leadership Team, managers participate in the co-adaptation of TIPS to their site and could be called upon to contribute to their site's monthly mentoring meetings. They will aid in the recruitment of therapists, parents, a therapist-champion, and a parent-partner for their site.
2. Therapists (n=600 with 50% anticipated response; n=300): PTs, OTs, SLPs providing outpatient pediatric rehabilitation services to children aged 0-12 years in each site, recruited via the managers and interested in utilizing FCT. Therapists will participate in the TIPS program, complete data collection instruments as prescribed, and aid in the recruitment of parents.
3. Parents (n=20/therapist with an anticipated response rate of 33%; n=2000 families per assessment time point): One-time data collection will be undertaken with two samples (one pre-, the other post-implementation) of parents or caregivers who received services (either in-person, virtually, or both) from at least one participating therapist in the previous 3 months.
4. Therapist-champion (n=20, one per site): Therapist selected based on their telehealth experience and on peer recognition within their organization. Therapist-champions are members of the Local Leadership Team participating in the co-adaptation of TIPS to their site and will oversee the monthly mentoring meetings.
5. Parent/patient-partner (n=20, one per site): Parent/patient-partners will primarily be recruited from family, parent or patient advisory committees at the participating sites or, in the absence of such initiatives, from regional, provincial, or national patient engagement programs. As members of the Local Leadership Team, parent/patient-partners participate in the co-adaptation of TIPS to their site and could be called upon to contribute to their site's monthly mentoring meetings.

Recruitment procedures will be flexible and will be adapted to the preferences, policies and procedures at each site. The recruitment of participants may be undertaken by email, sent directly to the potential participant by the research team (ex: therapists) or by the manager or therapist on behalf of the research team (e.g., parents).

Data collection Implementation data will be collected at least three times during each study period: pre-, per-, and post-implementation of TIPS. The additional data collection time point at 1 month per-TIPS will allow the documentation of the short-term impact of TIPS. Statistical analysis models will account for the inequivalent time intervals across study periods. A pre-post design was chosen to measure the intervention effectiveness outcomes and costs, using easily accessible service indicators and questionnaires administered to parents (obj. 4 + obj. 5), as per Type 3 hybrid designs. Qualitative data will be collected during (i.e., recording of monthly local mentoring meetings, and other meetings (as deemed appropriate by the therapist champion), in the vCoP discussions (as threads) and after (i.e., interviews with managers, therapist-champions, therapists and families) the implementation of TIPS.

Sample size justification Number of sites: A total of 20 sites across 8 Canadian provinces (grouped in 6 regions for the roll out of the intervention) are included in the study. Whenever possible, at least 3 sites per province were included to ensure sample diversity and enable the exploration of the provincial health systems' effects on the outcomes as well as to estimate site-related variations in outcomes. Five regions will include sites in the same province, while one region will consist of sites from 3 provinces where only one rehabilitation program was available.

Number of therapists: At the therapist level, implementation outcomes will be assessed 3 times during each period (pre-, per-, and post-TIPS implementation). Assuming an autocorrelation of repeated measures of r<0.3, data collected from 300 therapists will provide >80% power to detect moderate effect sizes (Cohen's d ≥ 0.5), employing a first-order autoregressive segmented regression model and a global type I error level of 5% accounting for multiplicity of outcome assessments (Sidak's correction).

Number of families: With a minimum expected sample size of 20 families per therapist being assessed pre- and/or post-TIPS implementation, statistical power will be >90% to detect even small effect-sizes (0.1< Cohen's d < 0.3) for the effectiveness outcomes i.e., change in wait times and change in families' perceptions of service quality.

Data analysis To evaluate the implementation (obj. 1), longitudinal mixed modeling accounting for and considering potential methodological issues associated with ITS analysis (e.g., auto-correlation, time-varying confounders) will be used to analyse implementation indicators (i.e., ADOPT-VR (Assessing Determinants of Prospective Take-up of Virtual Reality), therapists' self-reported FCT frequency, FCT fidelity self-perceived checklist, PRIME-SP). Changes will be documented short term (i.e., one month after the introduction of the TIPS) and long term (i.e., at the end of the TIPS, 12 months after its introduction). Models will be covariate-adjusted to reduce potential confounding bias, including the therapists' characteristics (e.g., gender, years of experience) and site characteristics (e.g., service provided, geography, general patients characteristics) to estimate associations of key explanatory variables alongside TIPS. Secondary analyses will explore heterogeneity in changes of outcome measures across genders, sites, therapists, and health jurisdiction levels.

To document site-specific co-adaptations of TIPS (obj. 2), proposed adaptations and decisions made by Local Leadership Team committee members will be documented during the discussion group in real-time on the logic model and in the TIPS training materials.

To identify factors influencing adoption and fidelity (obj. 3), recordings of monthly therapists' meetings, potential meetings between KBs and therapist champions) will be analyzed thematically, using a deductive-inductive approach guided by the Consolidated Framework for Implementation Research (CFIR) domains. Guided by an exploratory mixed methods approach, qualitative findings will be integrated with quantitative questionnaire results to further detail inferences.

To evaluate effectiveness (obj. 4) via estimated change in wait times (pre vs post), the confounder-adjusted analysis using generalized linear mixed effect models (GLMM) will employ a log-link function to account for the typically right-skewed nature of time data. Estimated fixed (intervention) effects for the effectiveness outcomes will be reported with Sidak-corrected 95% confidence intervals. To evaluate effectiveness via MPOC-20 (Measure of Process of Care - 20 questions) data, GLMM with nested random effects (families within therapists within sites) will be employed to control for the correlated nature of the data (i.e., the possibility that families have responded once or twice to the MPOC-20) and to account for therapist and site cluster effects. Analyses will be conducted for each of the five MPOC-20 domains and controlled for the same confounding variables described in the analysis for objective 1, as well as for family level variables (e.g., sociocultural background, child's age and gender).

Video-recorded interview data from therapists, managers, and parents will be analysed thematically using an inductive approach to better understand the breadth and depth of changes to pediatric rehabilitation service delivery, according to various stakeholder perspectives. Integration of quantitative and qualitative data using the aforementioned explanatory approach will allow us to uncover the plethora of effects of FCT on pediatric rehabilitation service delivery.

Total system costs related to the implementation of the TIPS, as well as the costs per participating therapist and per site, accounting for different organizational characteristics, will be calculated. Relative cost, an estimation of costs per client seen by therapist, and incremental ratios (i.e., change in costs to use the TIPS divided by change in the primary implementation indicators and secondary effectiveness outcomes) will also be calculated. Finally, societal costs, including families' costs and savings, will also be computed.

Ethical considerations The research ethics committees overseeing the 20 participating sites will approve this research project and be informed of any potential revisions of the protocol. Informed consent will be sought prior to data collection from participating managers, therapists, and parents. Participants will be assigned a unique identification number for denominalization purposes. Whenever posting content to the vCoP, therapists will be encouraged to use their name to promote open exchanges on the platform, but all users will also have the option of using a pseudonym if they prefer. The implementation of the TIPS (e.g., training, meetings) and all data collection (surveys, vCoP, interviews) will take place entirely online. Secure data collection and management solutions (e.g., REDCap, PIERCE) will be used to collect and store study data on institutional servers.

The implementation of TIPS will be gradual across regions, thus ensuring that the sites within the region are ready to participate in the project, taking into consideration institutional challenges such as availability of personnel or timeliness of the implementation of new telehealth modalities. Participants will be informed that study data will not constitute an evaluation of their professional performance. Some concerns are present in the literature that telehealth could increase health inequity and that wealthier families might benefit more from it. This project aims to support the use of FCT interventions with all Canadians families with a child with, or at risk of disability, while considering the interactions between personal, socio-economic, and cultural characteristics, as recommended. The team delivering TIPS is fully bilingual. TIPS and the study's data collection will be available in Canada's two official languages. A pre- and per-implementation consultation process will also be undertaken with First Nations Elders in order to take into account the needs of indigenous communities when delivering TIPS.

KNOWLEDGE TRANSFER In addition to the Local Leadership Team and the support provided to therapist champions, patient-oriented principles will be used within an integrated knowledge translation (iKT) approach to collaborate with knowledge users throughout the research process in order to inform research decisions. Specifically, four members of the research team (two parent-partner and two rehabilitation managers) have specifically been involved as knowledge users, and will be part of the study's Steering Committee. Principles for engaging with non-researchers in research will be respected (e.g., reviewing mutual expectations, providing meeting flexibility and clarification opportunities). The impact of the iKT approach will be assessed, using patient and organizational engagement criteria. Expected knowledge translation strategies include the presentation of study and site-specific data via a webinar for each participating site, as well as the publication of study findings via peer-reviewed publications and via public-facing publications on the research team's and project partners' websites, social media, and newsletters.

EXPECTED OUTCOMES This study will generate knowledge about how to implement family-centred telehealth and rehabilitation practices, inclusive of all families of children with, or at risk of, disability. The knowledge will be contextualized to support therapists working in varied settings and will contribute to building local capacity to sustain the use of FCT interventions. All training materials will be available across Canada and beyond. By increasing therapists' ability to provide telehealth services, the investigators hope to contribute to the transformation of pediatric rehabilitation service delivery, improve access to services, and foster greater well-being for families of children with, or at risk of, disability.

ELIGIBILITY:
Inclusion/Exclusion Criteria:

Managers:

* Person responsible for rehabilitation services at the site, or their delegate

Therapists:

* PTs, OTs, SLPs providing outpatient pediatric rehabilitation services to children aged 0-12 years in each site, recruited via the managers and interested in utilizing FCT

Parents:

* Parents or caregivers who received services (either in-person, virtually, or both) from at least one participating therapist in the previous 3 months

Therapist champion:

* Therapist selected based on their telehealth experience and on peer recognition within their organization.

Parent/patient-partners:

* Recruited from family, parent or patient advisory committees at the participating sites or, in the absence of such initiatives, from regional, provincial, or national patient engagement programs.

All:

* Can speak French or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2360 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
TIPS Therapist Survey-1 | 3 months prior to TIPS implementation
  The TIPS Therapist Survey contains sociodemographic information about the study participant (e.g., discipline, site, province, age), as well as the Therapists' Implementation Questionnaire (TIQ). The TIQ includes the ACCEPT-VFCC (Assessment of Competencies and Contributors to Enhance Practice Transition to Virtual Family Centred Care), a newly created tool inspired by the ADOPT-VR, yet specifically designed for telerehabilitation, the Family Centered Telerehabilitation (FCT) fidelity self-perceived checklist and the PRIME-SP (Pediatric Rehabilitation Intervention Measure of Engagement - Service Provider version).
TIPS Therapist Survey-2 | 2 months prior to TIPS implementation
  The TIPS Therapist Survey contains sociodemographic information about the study participant (e.g., discipline, site, province, age), as well as the Therapists' Implementation Questionnaire (TIQ). The TIQ includes the ACCEPT-VFCC (Assessment of Competencies and Contributors to Enhance Practice Transition to Virtual Family Centred Care), a newly created tool inspired by the ADOPT-VR, yet specifically designed for telerehabilitation, the Family Centered Telerehabilitation (FCT) fidelity self-perceived checklist and the PRIME-SP (Pediatric Rehabilitation Intervention Measure of Engagement - Service Provider version).
TIPS Therapist Survey-3 | 1 month prior to TIPS implementation
  The TIPS Therapist Survey contains sociodemographic information about the study participant (e.g., discipline, site, province, age), as well as the Therapists' Implementation Questionnaire (TIQ). The TIQ includes the ACCEPT-VFCC (Assessment of Competencies and Contributors to Enhance Practice Transition to Virtual Family Centred Care), a newly created tool inspired by the ADOPT-VR, yet specifically designed for telerehabilitation, the Family Centered Telerehabilitation (FCT) fidelity self-perceived checklist and the PRIME-SP (Pediatric Rehabilitation Intervention Measure of Engagement - Service Provider version).
TIPS Therapist Survey-4 | on day 1 of TIPS implementation
  The TIPS Therapist Survey contains sociodemographic information about the study participant (e.g., discipline, site, province, age), as well as the Therapists' Implementation Questionnaire (TIQ). The TIQ includes the ACCEPT-VFCC (Assessment of Competencies and Contributors to Enhance Practice Transition to Virtual Family Centred Care), a newly created tool inspired by the ADOPT-VR, yet specifically designed for telerehabilitation, the Family Centered Telerehabilitation (FCT) fidelity self-perceived checklist and the PRIME-SP (Pediatric Rehabilitation Intervention Measure of Engagement - Service Provider version).
TIPS Therapist Survey-5 | 1 month post TIPS commencement
  The TIPS Therapist Survey contains sociodemographic information about the study participant (e.g., discipline, site, province, age), as well as the Therapists' Implementation Questionnaire (TIQ). The TIQ includes the ACCEPT-VFCC (Assessment of Competencies and Contributors to Enhance Practice Transition to Virtual Family Centred Care), a newly created tool inspired by the ADOPT-VR, yet specifically designed for telerehabilitation, the Family Centered Telerehabilitation (FCT) fidelity self-perceived checklist and the PRIME-SP (Pediatric Rehabilitation Intervention Measure of Engagement - Service Provider version).
TIPS Therapist Survey-6 | 4 months post TIPS commencement
  The TIPS Therapist Survey contains sociodemographic information about the study participant (e.g., discipline, site, province, age), as well as the Therapists' Implementation Questionnaire (TIQ). The TIQ includes the ACCEPT-VFCC (Assessment of Competencies and Contributors to Enhance Practice Transition to Virtual Family Centred Care), a newly created tool inspired by the ADOPT-VR, yet specifically designed for telerehabilitation, the Family Centered Telerehabilitation (FCT) fidelity self-perceived checklist and the PRIME-SP (Pediatric Rehabilitation Intervention Measure of Engagement - Service Provider version).
TIPS Therapist Survey-7 | 8 months post TIPS commencement
  The TIPS Therapist Survey contains sociodemographic information about the study participant (e.g., discipline, site, province, age), as well as the Therapists' Implementation Questionnaire (TIQ). The TIQ includes the ACCEPT-VFCC (Assessment of Competencies and Contributors to Enhance Practice Transition to Virtual Family Centred Care), a newly created tool inspired by the ADOPT-VR, yet specifically designed for telerehabilitation, the Family Centered Telerehabilitation (FCT) fidelity self-perceived checklist and the PRIME-SP (Pediatric Rehabilitation Intervention Measure of Engagement - Service Provider version).
TIPS Therapist Survey-8 | 12 months post TIPS commencement
  The TIPS Therapist Survey contains sociodemographic information about the study participant (e.g., discipline, site, province, age), as well as the Therapists' Implementation Questionnaire (TIQ). The TIQ includes the ACCEPT-VFCC (Assessment of Competencies and Contributors to Enhance Practice Transition to Virtual Family Centred Care), a newly created tool inspired by the ADOPT-VR, yet specifically designed for telerehabilitation, the Family Centered Telerehabilitation (FCT) fidelity self-perceived checklist and the PRIME-SP (Pediatric Rehabilitation Intervention Measure of Engagement - Service Provider version).
TIPS Therapist Survey-9 | 3 months following the end of TIPS implementation
  The TIPS Therapist Survey contains sociodemographic information about the study participant (e.g., discipline, site, province, age), as well as the Therapists' Implementation Questionnaire (TIQ). The TIQ includes the ACCEPT-VFCC (Assessment of Competencies and Contributors to Enhance Practice Transition to Virtual Family Centred Care), a newly created tool inspired by the ADOPT-VR, yet specifically designed for telerehabilitation, the Family Centered Telerehabilitation (FCT) fidelity self-perceived checklist and the PRIME-SP (Pediatric Rehabilitation Intervention Measure of Engagement - Service Provider version).
TIPS Therapist Survey-10 | 6 months following the end of TIPS implementation
  The TIPS Therapist Survey contains sociodemographic information about the study participant (e.g., discipline, site, province, age), as well as the Therapists' Implementation Questionnaire (TIQ). The TIQ includes the ACCEPT-VFCC (Assessment of Competencies and Contributors to Enhance Practice Transition to Virtual Family Centred Care), a newly created tool inspired by the ADOPT-VR, yet specifically designed for telerehabilitation, the Family Centered Telerehabilitation (FCT) fidelity self-perceived checklist and the PRIME-SP (Pediatric Rehabilitation Intervention Measure of Engagement - Service Provider version).
TIPS Manager Survey (Pre-Implementation)-1 | 3 months prior to the commencement of TIPS implementation
  This survey includes sociodemographic information about the manager (e.g., academic degree, discipline, years of experience), the site profile (SPQ) which includes characteristics about the services provided, the organizations e-readiness, and service wait-time indicators.
TIPS Manager Survey (Pre-Implementation)-2 | on day 1 of TIPS implementation
  This survey includes sociodemographic information about the manager (e.g., academic degree, discipline, years of experience), the site profile (SPQ) which includes characteristics about the services provided, the organizations e-readiness, and service wait-time indicators.
TIPS Manager Survey (Post-Implementation) | within 6 months following the end of TIPS implementation
  This survey includes sociodemographic information about the manager (e.g., academic degree, discipline, years of experience), the site profile (SPQ) which includes characteristics about the services provided, the organizational e-readiness, service wait-time indicators, as well as the addition of organizational costs.
TIPS Therapist Champion Survey | once, 2 months prior to TIPS implementation
  This one-time survey is limited to the participant's sociodemographic information (e.g., discipline, years of experience), as well as their telerehabilitation experience, expertise, and training.
TIPS Parent Survey-1 | once, prior to day 1 of TIPS implementation
  This questionnaire contains The Family Questionnaire (Fam-Q) which collects sociodemographic information about the parent participants and their family (e.g., age, household income, family structure, remoteness) and the family costs and savings associated with accessing rehabilitation services, as well as the MPOC-20 (Measure of Process of Care - 20 questions).
TIPS Parent Survey-2 | once, within 6 months of the end of TIPS implementation
  This questionnaire contains The Family Questionnaire (Fam-Q) which collects sociodemographic information about the parent participants and their family (e.g., age, household income, family structure, remoteness) and the family costs and savings associated with accessing rehabilitation services, as well as the MPOC-20 (Measure of Process of Care - 20 questions).
TIPS Parent Partner Survey | once, 2 months prior to TIPS implementation
  This one-time survey is limited to the participant's sociodemographic characteristics (e.g., age, household income), their comfort level with technology, and their experiences with the site and the various service options (including telerehabilitation)
Semi-Structured Interviews | within 6 months following the end of TIPS implementation
  To explore all changes in service delivery (both negative and positive), stakeholders will be invited to participate in a video-recorded semi-structured interview post-implementation. The samples will include all managers, a sample of therapists (all local site champions and a subsample of therapists showing high or low adoption in different sites); and parents with diverse sociocultural characteristics and levels of perception of quality of care and experience with FCT. Parent, manager, therapist and therapist champion interviews will all be conducted only once with each participant.

SECONDARY OUTCOMES:
TIPS Logic Model | within 2 months prior to commencement of TIPS implementation
  A TIPS logic model will be developed by the research team based on best evidence to address FCT needs identified by therapists in a national survey and those recently reported by pediatric therapists in the literature and presented to the Local Leadership Team members for feedback. A discussion group format will be used to gather the Local Leadership Team members' input on site-specific TIPS co-adaptation (i.e., logic model, training materials). To document the Local Leadership Team members' characteristics (e.g., years of experience) and expertise (e.g., involvement and experience with telehealth services), they will be asked to complete a sociodemographic questionnaire prior to the discussion group.
Monthly therapist mentoring meetings | recorded at the frequency at which they occur (i.e., monthly) throughout the 11-months of the study in which they are scheduled
  Recordings of local monthly therapists' meetings, along with the vCoP discussion threads will be used to identify factors influencing therapists' intention to adopt and use FCT, site FCT implementation challenges and successes, and will facilitate better understanding of the impact of TIPS on clinical practice changes.
Virtual community of practice discussion threads and posts | collected regularly (i.e. monthly) over the 11 months of the support program
  Virtual community of practice discussion threads, along with recordings of local monthly therapists' meetings, will be used to identify factors influencing therapists' intention to adopt and use FCT, site FCT implementation challenges and successes, and will facilitate better understanding of the impact of TIPS on clinical practice changes.

CONTACTS AND LOCATIONS:
Overall Officials: Chantal Camden, PhD, Principal Investigator — École de réadaptation, CRCHUS, Université de Sherbrooke
Locations (3):
- Canada (3):
  - Centre intégré universitaire de santé et de services sociaux du Saguenay-Lac-Saint-Jean, Chicoutimi, Quebec
  - Centre intégré universitaire de santé et des services sociaux de l'Estrie - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec
  - Centre intégré universitaire de santé et de services sociaux de la Mauricie-et-du-Centre-du-Québec, Trois-Rivières, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hurtubise K, Gaboury I, Berbari J, Battista MC, Schuster T, Phoenix M, Rosenbaum P, Kraus De Camargo O, Lovo S, Pritchard-Wiart L, Zwicker JG, Beaudoin AJ, Morin M, Poder T, Gagnon MP, Roch G, Levac D, Tousignant M, Colquhoun H, Miller K, Churchill J, Robeson P, Ruegg A, Nault M, Camden C. Training Intervention and Program of Support for Fostering the Adoption of Family-Centered Telehealth in Pediatric Rehabilitation: Protocol for a Multimethod, Prospective, Hybrid Type 3 Implementation-Effectiveness Study. JMIR Res Protoc. 2022 Oct 28;11(10):e40218. doi: 10.2196/40218. PMID 36306158